CLINICAL TRIAL: NCT04532229
Title: A Multicenter, Prospective, Open and Single Arm Clinical Study of Nimotuzumab Combined With Concurrent Radiochemotherapy in the Treatment of Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG) in Children
Brief Title: Nimotuzumab in Combined With Chemoradiotherapy to Treat the Newly Diagnosed Diffuse Intrinsic Pontine Glioma in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-Nim-DIPG-1
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: Nimotuzumab; Temozolomide; DIPG
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Nimotuzumab+CRT(concurrent IMRT and TMZ)
  Interventions: Drug: Nimotuzumab+CRT(concurrent IMRT and TMZ)

INTERVENTIONS:
Drug: Nimotuzumab+CRT(concurrent IMRT and TMZ) — Drug: Nimotuzumab Concurrent radiochemotherapy period, 150mg/m2, weekly, for 6 weeks; Maintenance period, from the 7th to the 52nd week, 150mg/m2, every two weeks until disease progression or intolerable toxicity.
  Other Names: h-R3
  Drug: Temozolomide Concurrent radiochemotherapy period, 75mg/m2, daily, for 6 weeks; Maintenance period, rest from the 7th to 10th weeks, from the 11th week, 150-200mg/m2, day1 to day5, 21 days for a cycle, for 6 cycles.
  Other Names: TMZ
  Other Names: h-R3

SUMMARY:
This is a prospective, open-label, single arm, multicenter clinical study. The purpose of the study is to evaluate the clinical efficacy and safety of combination Nimotuzumab with concurrent radiochemotherapy in children with newly diagnosed diffuse intrinsic pontine glioma(DIPG).

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, open-label, single arm, multicenter study to evaluate the clinical efficacy and safety of combination Nimotuzumab with concurrent radiochemotherapy in children with newly diagnosed diffuse intrinsic pontine glioma(DIPG). The main endpoint is objective response rate, 1-year overall survival rate is also observed.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and sign a consent form;
2. Age 3-15 years old, gender unlimited;
3. Histology or imaging diagnosed as diffuse intrinsic pontine glioma, patients haven't received any anti-tumor treatment;
4. According to the RANO criteria, at least one measurable lesion;
5. Before enrollment, the results of laboratory examination are in accordance with:

   Blood routine test: platelet count ≥ 100 × 10^9/L; absolute neutrophil count ≥ 1.5 × 10^9/L or leukocyte count ≥ 3.0 × 10^9/L; hemoglobin ≥ 90g/L; Blood biochemistry: aspartate aminotransferase#AST# ≤ 3 ×Upper Limit Of Normal#ULN#; alanine aminotransferase#ALT# ≤ 3 × ULN; total bilirubin ≤ 1.5 × ULN; serum creatinine ≤ 1.5 × ULN;
6. Lansky score ≥ 60;
7. Expected survival time ≥ 3 months;
8. Fertile subjects are willing to take contraceptive measures during the study period.

Exclusion Criteria:

1. Recurrent DIPG;
2. Have received any other anti-tumor treatment for DIPG, including surgical treatment (except biopsy), chemotherapy, radiotherapy, targeted drugs, immunotherapy, etc;
3. Uncontrollable infection, epilepsy and / or hypertension and / or hyperglycemia;
4. Human immunodeficiency virus #HIV# infection or active hepatitis B infection or hepatitis C infection;
5. Active hemorrhage found by CT or MRI before inclusion and / or inability to carry out CT and MRI examination;
6. Major operation (except biopsy) were performed within four weeks before inclusion;
7. Decompensated heart failure (NYHA grades III and IV), unstable angina, acute myocardial infarction, persistent and clinically significant arrhythmia within three months of inclusion;
8. Have other malignant tumor history;
9. Known allergy to Nimotuzumab, temozolomide or its analogues or any component of the prescription;
10. Unable to tolerate radiotherapy;
11. Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2023-10-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate #ORR# assessed by the Independent Review Committee | Up to 12 months
  Proportion of patients with partial or complete response in tumor burden as defined by RECIST.

SECONDARY OUTCOMES:
1-year overall survival | Up to 12 months
  The possibility that a patient who has lived for 1 year after treatment will still survive. OS is defined as the time from enrollment to death.
Progression-free survival#PFS# | Up to 12 months
  PFS is defined as the time from enrollment to disease progression or death from any cause.
Incidence of adverse events | Up to 30 days after last administration of Nimotuzumab
  An adverse event is any adverse event that occurs in a patient or subject of a drug clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Yuan, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Xiaoguang Qiu, Study Chair — Beijing Tiantan Hospital
Locations (8):
- China (8):
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Xiangya Hospital of Centre-south University, Changsha, Hunan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Shandong Cancer Hospital, Jinan
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No